CLINICAL TRIAL: NCT00181870
Title: Open-Label Study of Equetro for the Treatment of Mania in Children Ages 6-12 With Bipolar I, Bipolar II, and Bipolar Spectrum Disorder
Brief Title: Equetro for the Treatment of Mania in Children Ages 6-12 With Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Shire (Industry)
Responsible Party: Janet Wozniak, MD, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-P-000763
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Bipolar Disorder; Mania
Keywords: bipolar disorder; children; mania; Equetro
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — Carbamazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: carbamazepine ER (Equetro)

SUMMARY:
This is an open-label pilot study of up to 1200 mg/day of carbamazepine ER (Equetro) in the treatment of children who meet DSM-IV criteria for Bipolar I, Bipolar II, or Bipolar Spectrum Disorder. The main goal of this study is to begin to address the void of information on safety, tolerability and effectiveness of Equetro in the treatment of Pediatric Bipolar Disorder.

DETAILED DESCRIPTION:
Initial clinical evidence suggests that carbamazepine (CBZ) may play a therapeutic role in the management of pediatric bipolar disorder. A recent study found that nearly 50% of patients taking immediate-release CBZ had side effects while only 20% of patients had side-effects after switching to an extended release (ER) version of the drug, despite high doses. In addition, with an ER formulation of CBZ there is a potential for decrease in peak-related side effects and improved efficacy with higher blood levels. Thus, an ER formulation of CBZ may improve effectiveness and adherence to treatment.

The goal of this pilot study is to evaluate the safety and effectiveness of Equetro in the treatment of bipolar I, bipolar II, and bipolar spectrum disorder in children ages 6-12 over the course of 8-weeks. We propose that during this exploratory study there will be sufficient safety, tolerability, and effectiveness of Equetro in the treatment of Pediatric Bipolar Disorder. The results of this study will be used to generate hypotheses for a larger randomized controlled clinical trial with explicit hypotheses and sufficient statistical power.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 6-12 years of age.
2. Subjects must have a DSM-IV diagnosis of bipolar I, bipolar II disorder or bipolar spectrum disorder and currently displaying manic, hypomanic, or mixed symptoms (with or without psychotic features) according to the DSM-IV based on clinical assessment and structured diagnostic interview (Kidd Schedule of Affective Disorders and Schizophrenia Epidemiological Version)(Kaufman, Birmaher et al. 1997). Bipolar Spectrum Disorder (or sub-threshold bipolar disorder) is operationalized as having severe mood disturbance, which meets DSM-IV Criteria A for bipolar disorder but meet fewer elements in criteria B (only require 2 items for elation category and 3 for irritability).
3. Subjects and their legal representative must have a level of understanding sufficient to communicate intelligently with the investigator and study coordinator, and to cooperate with all tests and examinations required by the protocol.
4. Subjects and their legal representative must be considered reliable.
5. Each subject and his/her authorized legal representative must understand the nature of the study. The subject's authorized legal representative must sign an informed consent document and the subject must sign an informed assent document.
6. Subjects must have an initial score on the Y-MRS total score of at least 20.
7. Subject must be able to participate in mandatory blood draws.
8. Subject must be able to swallow pills.
9. Subjects with comorbid ADHD, ODD, CD, anxiety and depressive disorders will be allowed to participate in the study provided they do not meet for any of the exclusionary criteria.
10. For concomitant therapy used to treat ADHD, subjects must have been on a stable dose of the medication for 1 month prior to study enrollment. The dose of the ADHD therapy will not change throughout the duration of the study. Strattera will not be allowed.

Exclusion Criteria:

1. Investigator and his/her immediate family; defined as the investigator's spouse, parent, child, grandparent, or grandchild.
2. Serious, unstable illness including hepatic, renal, gastroenterological, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.
3. Uncorrected hypothyroidism or hyperthyroidism.
4. History of sensitivity to carbamazepine or known sensitivity to any of the tricyclic compounds such as amitriptyline, desipramine, imipramine, protriptyline and nortriptyline. Severe allergies or multiple adverse drug reactions.
5. Non-febrile seizures without a clear and resolved etiology.
6. History of previous bone marrow depression
7. DSM-IV substance (except nicotine or caffeine) dependence within past 6 months.
8. Judged clinically to be at serious suicidal risk.
9. Any other concomitant medication with primarily central nervous system activity other than specified in Concomitant Medication portion of the protocol.
10. A non-responder or a history of intolerance to carbamazepine on an adequate trial (2 months or more at an adequate dose) as determined by the clinician.
11. Current diagnosis of schizophrenia.
12. Pregnant or nursing females.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2005-07; Primary Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
symptom reduction measured by YMRS | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Janet Wozniak, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States